CLINICAL TRIAL: NCT03856892
Title: Breath, Stress and Health: a Biocultural Study of Hatha Yoga Practice
Acronym: Yoga
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Carol Worthman, Professor of Anthropology, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00107267
Record Dates: First submitted 2019-02-26; First posted 2019-02-27 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Stress, Physiological; Stress, Psychological
Keywords: Yoga; Breath-based yoga; Stress management; Meditation; Hatha yoga; Anxiety mitigation; Mental health; Longevity
MeSH Terms: conditions — Stress, Psychological; Psychological Well-Being | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active Study Group (Experimental): Participants randomized to the Active Study Group are asked to follow a daily routine of the three protocols of psycho-physical yoga component techniques: Slow Engaged Dynamic Asana (SEDA), Breath Regulated Engaged Meditation (BREM), Sound Heart Engaged Meditation (SHEM). This intervention involves more hours in daily practice to equate to a "high dose" of breath and meditative techniques.
  Interventions: Other: High Dose Yoga
- Active Control (Active Comparator): Participants randomized to the Active Control study arm are asked to follow a daily routine of low-to mid-intensity body posture practice that is body-based and has minimal breath or meditative elements. This intervention involves fewer hours in daily practice to equate to a "medium dose" of body focused techniques
  Interventions: Other: Medium Dose Yoga
- Passive Control (No Intervention): Participants randomized to the Passive Control study arm do not receive a study intervention.

INTERVENTIONS:
Other: High Dose Yoga — Participants engage in an intensive full yoga practice of hatha breath-based practices and inner meditative techniques along with body-based asana. Intensive level uses breath, management of abdomen, inner focus in all practices. The "high dose" of yoga is an interpretation of the Translational Model of Yoga (TMY) and Yoga Process formula, both developed in this study's cultural research: a systematized psycho-physical yoga method of Hatha Zone (HZ) focus (below-navel, exhale, inner focus), incorporating key components of practice-focus-surrender (PFS) approach and repeat-engage-trust (RET) elements.
  Arms: Active Study Group
Other: Medium Dose Yoga — The "medium dose" of yoga is a regular practice of primarily body-posture training with minimal reference to the breath, but with a longer period of time duration in training prior to intervention commencement. Participants have 5 months of pre-training before initiating the intervention.
  Arms: Active Control

SUMMARY:
This study aims to contribute uniquely to stress, longevity, and mental health research in two ways: by identifying clear protocols of breath-based yoga-meditative practice based on original materials; that are subsequently assessed with established scientific stress, biochemical immunity and longevity markers, and validated psychological measures that relate to mental health.

DETAILED DESCRIPTION:
This study aims to contribute uniquely to stress, longevity, and mental health research in two ways: by identifying clear protocols of breath-based yoga-meditative practice based on original materials; that are subsequently assessed with established scientific stress markers across the sympathetic-adreno-medullar (SAM) axis, biochemical immunity and longevity markers, and validated psychological measures as related to mental health. The study couples emic perspectives from the traditional yoga knowledge base, both textual and practice, with empirical measures from science as an opportunity to bridge these worlds as a first known study of hatha yoga to be tackled by the means and methods of biocultural anthropology. It therefore highlights the importance of context and detail in terms of assessing human behavioral practices, where accuracy in terms of definitions, technique detail, and original purported intentions and outcomes are addressed as relevant when measuring and explaining empirical outcomes under modern research mixed methods.

ELIGIBILITY:
Inclusion Criteria:

* Novice to breath-based yoga practice
* Multicultural international participant base
* Fluent in English comprehension and reading
* In general good health
* Have a smartphone or similar device in order to receive surveys on a dedicated app

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-09-17 (Actual)

PRIMARY OUTCOMES:
Change in Heart Rate Variability (HRV) Between Study Arms | Baseline, up to 6 months
  Heart rate variability (HRV) is measured by electrocardiogram.

SECONDARY OUTCOMES:
Change in Heart Rate Variability (HRV) Between High and Low Participation Level | Baseline, up to 6 months
  Heart rate variability (HRV) is measured by electrocardiogram. Participants will be categorized as higher teacher-rated "engaged participation" or lower teacher-rated "engaged participation" and these groups will be compared.
Change in Skin Conductance Level (SCL) Between Study Arms | Baseline, up to 6 months
  Skin conductance level (SCL) is measured by electrodermal activity (EDA).
Change in Skin conductance level (SCL) Between High and Low Participation Level | Baseline, up to 6 months
  Skin conductance level (SCL) is measured by electrodermal activity (EDA). Participants will be categorized as higher teacher-rated "engaged participation" or lower teacher-rated "engaged participation" and these groups will be compared.
Change in Skin Conductance Response Between Study Arms | Baseline, up to 6 months
  Skin conductance response is measured by electrodermal activity (EDA).
Change in Skin Conductance Response Between High and Low Participation Level | Baseline, up to 6 months
  Skin conductance response is measured by electrodermal activity (EDA). Participants will be categorized as higher teacher-rated "engaged participation" or lower teacher-rated "engaged participation" and these groups will be compared.
Change in Reactive Oxygen Species (ROS) Levels Between Study Arms | Baseline, up to 6 months
  Oxidative stress will be measured by ROS levels.
Change in Reactive Oxygen Species (ROS) Between High and Low Participation Level | Baseline, up to 6 months
  Oxidative stress will be measured by ROS levels. Participants will be categorized as higher teacher-rated "engaged participation" or lower teacher-rated "engaged participation" and these groups will be compared.
Change in Total Antioxidant Status (TAS) Between Study Arms | Baseline, up to 6 months
  Change in TAS will be measured by blood sample analysis.
Change in Total Antioxidant Status (TAS) Between High and Low Participation Level | Baseline, up to 6 months
  Change in TAS will be measured by blood sample analysis. Participants will be categorized as higher teacher-rated "engaged participation" or lower teacher-rated "engaged participation" and these groups will be compared.
Change in Levels of Antioxidant Enzyme Glutathione (GSH) Between Study Arms | Baseline, up to 6 months
  Glutathione (GSH) is an antioxidant capable of preventing damage to important cellular components caused by reactive oxygen species such as free radicals, peroxides, lipid peroxides, and heavy metals. Change in levels of GSH will be measured by blood sample analysis.
Change in levels of antioxidant enzyme Glutathione (GSH) Between High and Low Participation Level | Baseline, up to 6 months
  Glutathione (GSH) is an antioxidant capable of preventing damage to important cellular components caused by reactive oxygen species such as free radicals, peroxides, lipid peroxides, and heavy metals. Change in levels of GSH will be measured by blood sample analysis. Participants will be categorized as higher teacher-rated "engaged participation" or lower teacher-rated "engaged participation" and these groups will be compared.
Change in Levels of Circulating IL-6 Between Study Arms | Baseline, up to 6 months
  Interleukin 6 (IL-6) is an interleukin that acts as both a pro-inflammatory cytokine and an anti-inflammatory myokine. Levels of circulating IL-6 will be assessed by blood sample analysis.
Change in levels of circulating IL-6 Between High and Low Participation Level | Baseline, up to 6 months
  Interleukin 6 (IL-6) is an interleukin that acts as both a pro-inflammatory cytokine and an anti-inflammatory myokine. Levels of circulating IL-6 will be assessed by blood sample analysis. Participants will be categorized as higher teacher-rated "engaged participation" or lower teacher-rated "engaged participation" and these groups will be compared.
Change in Levels of Circulating Tumor-Necrosis Factor-alpha (TNF-α) Between Study Arms | Baseline, up to 6 months
  Tumor necrosis factor is a cell signaling protein (cytokine) involved in systemic inflammation. Change in levels of circulating TNF-α will be assessed by blood sample analysis.
Change in levels of circulating TNF-α Between High and Low Participation Level | Baseline, up to 6 months
  Tumor necrosis factor is a cell signaling protein (cytokine) involved in systemic inflammation. Change in levels of Circulating TNF-α will be assessed by blood sample analysis. Participants will be categorized as higher teacher-rated "engaged participation" or lower teacher-rated "engaged participation" and these groups will be compared.
Change in Upper Abdominal Muscle Tension Between Study Arms | Baseline, up to 6 months
  Upper abdominal muscular tension levels is assessed as Muscle Tone and Muscle Stiffness, and is measured by the MyotonPlus digital palpation device at a precise site on the upper region of the Rectus Abdominis (RA) muscle.
Change in Upper Abdominal Muscle Tension Between High and Low Participation Level | Baseline, up to 6 months
  Upper abdominal muscular tension levels is assessed as Muscle Tone and Muscle Stiffness, and is measured by the MyotonPlus digital palpation device at a precise site on the upper region of the Rectus Abdominis (RA) muscle.
Change in Self-assessment Questions Covering "how do you feel" score | Baseline, up to 6 months
  Self-assessment questions covering "how do you feel", with ongoing 3 daily-based questions once a week.
Change in Perceived Stress Reactivity Scale (PSRS) Score | Baseline, up to 6 months
  The Perceived Stress Reactivity Scale (PSRS), a 23-item questionnaire with 5 subscales (Prolonged Reactivity, Reactivity to Failure, Reactivity to Social Conflicts, Reactivity to Work Overload, and Reactivity to Social Evaluation) and 1 overall scale. The PSRS overall score ranges from 0 to 30 and higher scores are associated with increased symptoms of depression and sleep disturbances.
Change in Perceived Stress Scale (PSS) Score | Baseline, up to 6 months
  The Perceived Stress Scale (PSS) is a 10-item instrument assessing feelings and thoughts related to stress during the past month. Each item is rated on a 5-point scale ranging from never (0) to very often (4). Total scores range from 0 to 40 with higher scores indicating higher perceived stress.
Change in Difficulties in Emotion Regulation Scale (DERS) Score | Baseline, up to 6 months
  The Difficulties in Emotion Regulation Scale (DERS) is a 36-item instrument assessing emotion dysregulation and includes six subscales (non-acceptance of emotions, difficulty with goal-directed behavior in the presence of negative emotions, difficulty controlling impulses in the presence of negative emotions, lack of awareness of emotions, limited use of effective emotion regulation strategies, and lack of understanding of emotions). Responses are scaled from 1 (almost never) to 5 (almost always). Total raw scores range from 36 to 180; certain items are reverse scored so that higher scores indicate increased difficulty with emotion regulation.
Change in Depression Anxiety and Stress Scale (DASS) Score | Baseline, up to 6 months
  The DASS is a 42-item self-administered questionnaire designed to measure the magnitude of three negative emotional states: depression, anxiety, and stress. The DASS-Depression focuses on reports of low mood, motivation, and self-esteem, DASS-anxiety on physiological arousal, perceived panic, and fear, and DASS-stress on tension and irritability. Individual patient scores on the DASS subscales can be interpreted by converting them to z-scores and comparing to the normative values contained within the DASS manual. A z-score < 0.5 is considered to be within the normal range, a z-score of 0.5 to 1.0 is mild, 1.0 to 2.0 is moderate, 2.0 to 3.0 is considered severe, and z-scores > 3 are considered to be extremely severe depression/anxiety/stress.
Change in Penn State Worry Questionnaire (PSWQ) Score | Baseline, up to 6 months
  The Penn State Worry Questionnaire (PSWQ) is a self-administered, 16-item, Likert-type scale designed to measure the trait of worry. Responses to items are rated from 1 to 5 where less worry = 1 and a lot of worry = 5. Total scores range from 16 to 80 and higher scores indicate greater severity of the trait of worry.
Change in Positive and Negative Affect Scale (PANAS) Score | Baseline, up to 6 months
  The Positive and Negative Affect Scale (PANAS) consists of 10 positively and 10 negatively valanced word items. Items are rated by the participant for the extent they are feeling this "right now" on a scale of 1- slightly or not at all through 5- extremely. Total scores can range from 10 to 50, with higher scores representing higher levels of positive effect and lower scores having negative effect.
Change in Beck Depression Inventory (BDI-II) Score | Baseline, up to 6 months
  The BDI-II is a self-report 21-item scale used to assess the current severity of depression. Each item is rated on a four-point scale (0 to 3) with possible total scores ranging from 0 to 63. Scores provide a measure of the severity of self-reported depression: 0 -9 minimal, 10 -16 mild, 17-29 moderate, and 30 - 63 severe.
Change in Beck Anxiety Inventory (BAI-II) Score | Baseline, up to 6 months
  The BAI-II is a 21-item self-report measure of anxiety symptoms, rated on a 4-point Likert scale. Items are rated from 0 = not at all to 3 = severely. Total scores range from 0 to 63 and higher scores indicate greater anxiety.
Change in Profile of Mood States (POMS) Score | Baseline, up to 6 months
  The Profile of Mood States (POMS) scale is a 30-item psychological rating scale used to assess transient, distinct mood states. Participants rate the extent to which they feel unhappy, blue, lonely, gloomy, and worthless on a scale from 0 (not at all) to 4 (extremely). Scores range from 0 to 120 with higher scores reflecting a more negative mood state.
Change in Coping Self-efficacy Scale (CSES) Score | Baseline, up to 6 months
  The CSES is a 26-item scale that measures one's perceived ability to cope with life's difficulties. Responses are given on a scale from 0 to 10 where 0 = cannot do at all and 10 = certain can do. Total scores range from 0 to 260 where higher scores indicate greater self-efficacy with coping skills.
Changes in Multidimensional Assessment of Interoceptive Awareness (MAIA) 8-Subscale Scores | Baseline, up to 6 months
  The Multidimensional Assessment of Interoceptive Awareness (MAIA) assesses various aspects of interoception with 8 subscales of: Noticing, Not-Distracting, Not-Worrying, Attention Regulation, Emotional Awareness, Self-Regulation, Body Listening, and Trusting. The subscales include 3 to 7 items and scored by taking the average of the item responses. Responses are given on a 6-point scale where "never" = 0 and "always" = 5. Total scores for each subscale range from 0 to 5 and higher scores indicate greater levels of interoceptive awareness.
Change in Mindful Attention Awareness Scale (MAAS) Score | Baseline, up to 6 months
  The Mindful Attention Awareness Scale (MAAS) is a 15-item instrument assessing mindfulness (attention to what is occurring in the present). Responses are given on a 6-point scale where "almost always" = 1 and "almost never" = 6. The total score is the average of responses to the 15 items and ranges from 1 to 6 where higher scores indicate greater mindfulness to the present moment.
Change in Compassion Scale (CS) Score | Baseline, up to 6 months
  The Compassion Scale (CS) is a 16-item instrument assessing compassion for others. Responses are given on a 5-point scale where "almost never" = 1 and "almost always" = 5. The total score is the average of responses to the 16 items and ranges from 1 to 5 where higher scores indicate greater compassion towards others.
Change in Self-Compassion Scale - Short Form (SCS-SF) Score | Baseline, up to 6 months
  The Self-Compassion Scale - Short Form (SCS-SF) is a 12-item instrument assessing self-compassion. Responses are given on a 5-point scale where "almost never" = 1 and "almost always" = 5. The total score is the average of responses to the 12 items and ranges from 1 to 5 where higher scores indicate greater self-compassion.
Change in Five Facet Mindfulness Questionnaire (FFMQ) Score | Baseline, up to 6 months
  The Five Facet Mindfulness Questionnaire (FFMQ) is a 39-item instrument with five subscales of: Observing, Describing, Acting with Awareness, Nonjudging, and Nonreactivity. Responses are given on a 5-point scale where "never or very rarely true" = 1 and "very often or always true" = 5. Scores can be obtained for each subscale and for a total score by averaging item responses. Total scores range from 1 to 5 where higher scores indicate greater mindfulness.
Change in Heartland Forgiveness Scale Score | Baseline, up to 6 months
  The Heartland Forgiveness Scale is an 18-item instrument assessing dispositional forgiveness, with 3 subscales of: Forgiveness of Self, Forgiveness of Others, and Forgiveness of Situations. Responses are given on a 7-point scale where "almost always false of me" = 1 and "almost always true of me" = 7. Total scores for each subscale range from 6 to 42, and the overall total score ranges from 18 to 126. Higher scores indicate greater dispositional forgiveness.
Change in Cognitive and Affective Mindfulness Scale - Revised (CAMS-R) Score | Baseline, up to 6 months
  The Cognitive and Affective Mindfulness Scale- Revised (CAMS-R) instrument assessing mindfulness with 12 items. Responses are given on a 4-point scale where "rarely/not at all" = 1 and "almost always" = 5. The total score ranges from 12 to 48 and higher scores indicate greater mindfulness.
Change in Gratitude Questionnaire - Six Item Form (GQ-6) Score | Baseline, up to 6 months
  The Gratitude Questionnaire - Six Item Form (GQ-6) instrument measures the experience of gratitude in daily life with 6 items. Responses are given on a 7-point scale where "strongly disagree" = 1 and "strongly agree" = 7. The total score is the average of responses to the 6 items and ranges from 1 to 7 where higher scores indicate greater gratitude.
Change in Spiritual Meaning Scale (SMS) Score | Baseline, up to 6 months
  The Spiritual Meaning Scale (SMS) measures an individuals belief that life has a purpose, will, or way. The 14 items are rated on a 5-point Likert scale where "I totally disagree" = 1 and "I totally agree" = 5. Total scores range from 14 to 70 where higher scores indicate greater feelings of spiritual meaning.
Change in Telomere Length (TL) | Baseline, up to 6 months
  Telomeres are caps at the ends of chromosomes that, based on primary research, are shown to shorten each time a cell divides. Telomere length (TL) is used as is a marker of cellular aging as shorter telomeres indicate limited cellular life, an indicator of senescence, used overall to comment on longevity of those being measured. Population studies use telomere length (TL) in studies of population health and lifespan. Telomere length (TL) will be measured by blood sample analysis.

OTHER OUTCOMES:
Change in Brain-derived Neurotrophic Factor (BDNF) Level in Blood Serum Between Study Arms | Baseline, up to 6 months
  Brain-derived neurotrophic factor is a member of the neurotrophin family of growth factors, will be measured by blood sample analysis.
Change in Growth Hormone Level in Blood Serum Between Study Arms | Baseline, up to 6 months
  Change in Growth Hormone level will be measured by blood sample analysis.
Change in Oxytocin Level in Blood Serum Between Study Arms | Baseline, up to 6 months
  Change in Oxytocin level will be measured by blood sample analysis.
Change in Ghrelin Level in Blood Serum Between Study Arms | Baseline, up to 6 months
  Change in Ghrelin level will be measured by blood sample analysis.
Change in Leptin Level in Blood Serum Between Study Arms | Baseline, up to 6 months
  Change in Leptin level will be measured by blood sample analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Dallaghan, PhD, Principal Investigator — Emory University
Locations (1):
- Kaivalyadhama Yoga Institute, Lonavla, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be made available for sharing with other researchers following deidentification.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available for sharing beginning immediately and ending 3 years after publication of the results from this study.
Access Criteria: Data will be available for sharing with researchers who provide a methodologically sound proposal, for the purposes of achieving the aims of the approved proposal. Proposals should be directed to paul.dallaghan@cuanschutz.edu. To gain access, requestors will need to sign a data access agreement.